CLINICAL TRIAL: NCT05797688
Title: Use of Autologous Adipose-derived Stem Cell to Treat Chronic Wounds
Brief Title: Adipose-derived Stem Cells to Treat Chronic Wounds.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Collaborators: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15586
Record Dates: First submitted 2016-12-23; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2016-12

CONDITIONS: Wound of Skin
Keywords: Chronic Wound; Chronic Ulcer; stem cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients will undergo a fat harvest procedure and the tissue will then be processed by The Celution System to isolate a 5 mL aliquot including stem cells. This will then be injected into the base and within in perimeter of the target wound.
  Interventions: Device: The Celution System

INTERVENTIONS:
Device: The Celution System — The Celution System will isolate regenerative cells, including stem cells, from fat harvested from the treatment patients.
  Other Names: Celution, Adipose-derived cell processor

SUMMARY:
The goal of this study is to determine whether autologous, adipose-derived regenerative cells improve the healing of chronic wounds. Ten patients will undergo fat harvest and peri-wound injection of the isolated cells in addition to the standard of care for the treatment of their chronic wound. Wound healing will be followed over 24 weeks.

DETAILED DESCRIPTION:
This study will be an open-label, preliminary, proof-of-concept trial. Ten patients will undergo debridement of their wound per the standard of care currently offered by Winthrop University Hospital along with concurrent fat harvest according to the standard protocols of the Winthrop University Hospital Plastic surgeons. The harvested fat will be immediately processed using an automated system to isolate regenerative cells, including stem cells. This will be followed by same-day subcutaneous injection of the isolated cells into the debrided wound site. The patients will then undergo weekly wound debridements according to the current standard of care treatment protocols. They will be followed weekly for 24 weeks in the outpatient wound clinic and observed for pain, erythema of the injection site, wound infection, edema, fever, bleeding and wound healing as measured by wound size and area. Fat harvest and subcutaneous injection will be repeated 3 months after the initial procedure if the wound has not decreased in size by at least 40%. Patients can undergo a maximum of 2 cycles of fat harvest and cell injection.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must agree to adhere to all protocol procedures and return for weekly scheduled wound assessment visits, including requirements for taking and abstaining from medications.
2. Subject is willing and able to read, understand and sign a written Informed Consent to participate in the study or have an appropriate representative available to do so.
3. Subject must have a full thickness Stage III or Stage IV pressure ulcer, deep venous ulcer, deep diabetic ulcer, ischemic ulcer, abdominal wound, nonhealing surgical site or sickle cell ulcer. For subjects with more than one wound that meet these criteria, the largest qualifying wound will be treated.
4. Subject has adequate (>200 mL) abdominal or other subcutaneous adipose tissue accessible by syringe-based fat harvest and is able to undergo a fat harvest procedure in the opinion of the investigator or per facility guidelines and has activated platelet thromboplastin time (aPTT) within the normal reference range at the time of the fat harvest procedure and no contraindication to fat harvest.
5. Subject's wound has been refractory to standard of care (no objective/measureable signs of healing) for at least 30 days.

Exclusion Criteria:

1. Subject has local infection with erythema > 2 cm, or involving structures deeper than skin and subcutaneous tissues (e.g., abscess, osteomyelitis, septic arthritis, fasciitis), or associated with local wound complications such as prosthetic materials or protruding surgical hardware.
2. Subject has ≥ 2 of the following signs of systemic inflammatory response syndrome (SIRS) or septic shock within 7 days of screening:

   * Temperature > 38°C or < 36°C
   * Heart rate > 90 beats/min
   * Respiratory rate > 20 breaths/min or PaCO2 < 32 mm Hg
   * White blood cell count > 12,000 or < 4,000 cells/μL or ≥ 10% immature (band) forms.
3. Subject has received biologic or cell therapy within 12 weeks of initiation of the study.
4. Subject not eligible for syringe-based liposuction of at least 200 mL of subcutaneous adipose tissue, including therapeutic anticoagulation with INR >1.7 or PTT >60, or receiving GIIb/IIIa inhibitors within 2 weeks prior to the study.
5. Subject has squamous cell carcinoma, basal cell carcinoma, melanoma or skin carcinoma of the affected limb or area and underwent treatment within the last year.
6. Subject is pregnant as determined by a positive pregnancy test prior to procedure, or breast-feeding.
7. Clinically significant abnormal findings on laboratory screening panels, including hemoglobin ≤10 g/dL.
8. Hepatic dysfunction, as defined as aspartate aminotransferase (AST), alanine aminotranferase (ALT), or bilirubin level > 1.5 times the upper limit of normal range (x ULN) prior to randomization.
9. Chronic renal insufficiency as defined as a serum creatinine > 2.0 mg/dL or requires dialysis.
10. History of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by weekly evalutation of the occurrence of wound infection, redness, swelling, pain, fever, chills, bleeding, and wound healing. | 1 year

SECONDARY OUTCOMES:
Complete wound healing | 1 year
  Wounds will be evaluated for 100% epithelialization with no drainage.
Time to healing | 1 year
  The time when complete healing occurs will be recorded, up to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Harold Brem, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: No